CLINICAL TRIAL: NCT02719951
Title: Glutaminergic Transmission in Autism : Molecular Imaging Exploration
Acronym: TANGAU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PRIA 14 FBB / TANGAU
Record Dates: First submitted 2016-03-09; First posted 2016-03-25 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Autism; Fragile-X Syndrome (FXS); Healthy Volunteers
Keywords: autism; fragile X syndrome (FXS); PET (Positron Emission Tomography); glutamate
MeSH Terms: conditions — Autistic Disorder; Fragile X Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- autistic patients (Experimental): [18F]FPEB PET imaging MRI (Magnetic Resonance Imaging) Biological samples
  Interventions: Drug: [18F]FPEB PET imaging; Other: Biological samples; Other: MRI
- FXS patients (Experimental): [18F]FPEB PET imaging MRI Biological samples
  Interventions: Drug: [18F]FPEB PET imaging; Other: Biological samples; Other: MRI
- Healthy subjects (Experimental): [18F]FPEB PET imaging MRI Biological samples
  Interventions: Drug: [18F]FPEB PET imaging; Other: Biological samples; Other: MRI

INTERVENTIONS:
Drug: [18F]FPEB PET imaging — PET exam
Other: Biological samples — blood sample and urine sample
Other: MRI — MRI exam

SUMMARY:
Glutamatergic transmission exploration using PET (Positron Emission Tomography) imaging in autism compared to Fragile-X Syndrome ( FXS) and Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Male
* Between 18 years-old and 45 years-old
* Informed, written consent obtained from patient or his representant
* Subject with an affiliation to French social security
* For autistic patient : patient with diagnosis of ASD (Autistic Spectrum Disorders) following DSM-IV or DSM-5 criteria with recommended tools (ADI-R and/or ADOS)
* For FXS patient : diagnosis of FXS and confirmation of total mutation of FMR1

Exclusion Criteria:

* Contraindications to MRI
* Excessive use of alcohol or drug, or addiction to alcohol or drug during last 6 months
* Any unstable or uncontrolled disease, clinically significant
* Participation to an other experimental protocol with drug or irradiant exam
* Person under exclusion period because of previous participation to an other experimental protocol
* Person under temporary guardianship
* Forbidden treatments : any psychotropic treatment for 4 last weeks before PET exam and changing durably glutaminergic transmission directly or undirectly
* For healthy subjects : adult under guardianship, medical history of central nervous system disease, medical history of attention deficit hyperactivity disorder, past or present psychiatric or neurologic disorder (MINI DSM-IV)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-04; Primary Completion 2018-11-15 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
cerebral glutaminergic activity assessed by binding potential of [18F]FPEB | An average of 3 years

SECONDARY OUTCOMES:
distribution volume of [18F]FPEB | An average of 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data.

REFERENCES:
- [Result] Dupont AC, Serriere S, Barantin L, Vercouillie J, Tauber C, Gissot V, Bodard S, Chicheri G, Chalon S, Bonnet-Brilhault PF, Santiago-Ribeiro PM, Arlicot N. Study of influence of the glutamatergic concentration of [18F]FPEB binding to metabotropic glutamate receptor subtype 5 with N-acetylcysteine challenge in rats and SRM/PET study in human healthy volunteers. Transl Psychiatry. 2021 Jan 20;11(1):66. doi: 10.1038/s41398-020-01152-2. PMID 33473111